CLINICAL TRIAL: NCT01110356
Title: A Multicentre Randomised Placebo-controlled Study to Assess the Efficacy and Safety of a Single Administration of Ferric Carboxymaltose in Improving Fatigue Symptoms in Iron-deficient Non-anaemic Women of Child Bearing Age
Brief Title: Ferric Carboxymaltose Treatment to Improve Fatigue Symptoms in Iron-deficient Non-anaemic Women of Child Bearing Age
Acronym: Prefer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vifor Pharma (Industry)
Collaborators: SGS S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: IDNA 2009-01
Record Dates: First submitted 2010-04-22; First posted 2010-04-26 (Estimated); Last update posted 2012-11-15 (Estimated); Status verified 2012-11

CONDITIONS: Iron Deficiency
MeSH Terms: conditions — Iron Deficiencies | interventions — ferric carboxymaltose; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ferinject (Experimental)
  Interventions: Drug: Ferinject
- Saline (Placebo Comparator)
  Interventions: Other: Saline

INTERVENTIONS:
Drug: Ferinject — Ferric carboxymaltose will be provided in 2 vials of 10 mL containing each 500 mg iron, which will be diluted in 250 mL normal saline for injection. Study drug will be administered by drip infusion immediately after preparation over a minimum of 15 minutes. Placebo patients will be administered 250 mL normal saline for injection over a minimum of 15 minutes.
  Arms: Ferinject
Other: Saline — Placebo patients will be administered 250 mL normal saline for intravenous drip over a minimum of 15 minutes.
  Arms: Saline

SUMMARY:
research study of Ferric carboxymaltose to treat fatigue/exhaustion symptoms, believed to be due to iron deficiency.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent prior to study specific procedures.
* Premenopausal, regularly menstruating women.
* Age ≥18 years.
* Body weight between 50 and 90 kg.
* Haemoglobin ≥115 g/L.
* Iron deficiency at screening defined as follows:
* S-ferritin level <50 ng/mL, AND, TfS <20%, OR,
* S-ferritin level <15 ng/mL.
* Serum C-reactive protein:
* <5 mg/L if not on oral contraception, OR,
* <20 mg/L if use of oral contraception.
* Minimum total score of 5 on the Piper Fatigue Scale (PFS) (mean of items 2 to 23).
* Negative pregnancy test (serum human chorionic gonadotropin (hCG) at screening.
* Normal levels of vitamin B12 and folic acid at screening.
* Adequate contraception during the study period and for 1 month following study completion.
* Availability and willingness to complete all study visits and procedures per protocol.

Exclusion Criteria:

* Haemoglobin level <115 g/L.
* Haemoglobinopathy.
* Haemochromatose.
* Major depressive disorder based on Patient Health Questionnaire (PHQ-9) (5 items with scores ≥2; one of which corresponds to question number 1 or 2).
* Any active or unstable concurrent medical condition (e.g., cancer, renal dysfunction, liver dysfunction (aspartate aminotransferase (AST); alanine aminotransferase (ALT) >3-fold upper limit), angina (Class IV).
* Known human immunodeficiency virus/acquired immunodeficiency syndrome, hepatitis B virus or hepatitis C virus infection.
* Chronic inflammatory disease (e.g., rheumatoid arthritis; inflammatory bowel disease).
* Documented history of clinically significant level of sleep apnoea defined as 5 or more episodes per hour of any type of apnoea.
* Intake of concurrent medications that could interfere with physical or mental performance (e.g., antidepressive, antihistamines, narcotic or any chemotherapeutic agents known to cause drowsiness).
* Important recent weight loss (>10% within the past month).
* Body weight <50 kg or >90 kg.
* Thyroid dysfunction, thyroid stimulating hormone >4 μU/mL.
* Intake of iron preparations 4 weeks prior to screening.
* Use of gestagens e.g., Implanon, Mirena, Depo-Provera for menstruation repression (see Section 7.7, Prohibited Therapy or Concomitant Treatment, page 35).
* Known hypersensitivity to FCM or to any other iron preparation.
* Pregnancy (positive hCG test at screening) or breast feeding.
* Participation in any other interventional trial within 4 weeks prior to screening.
* Inability to fully comprehend and/or perform study procedures or provide written consent in the Investigator's opinion.
* Subject is not using adequate contraceptive precautions during the study and for up to 1 month after the last dose of the study medication. A highly effective method of birth control is defined as those which result in a low failure rate (i.e., less than 1% per year) when used consistently and correctly such as implants, injectables, combined oral contraceptives, some intra-uterine devices, sexual abstinence or vasectomised partner.
* Subject previously has entered this study.
* Subject will not be available for follow-up assessments.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 294 (Actual)
Dates: Start 2010-06; Primary Completion 2011-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
To assess the efficacy of a single intravenous (IV) administration of FCM (1,000 mg) compared with placebo in improving fatigue symptoms in IDNA women of child bearing age. | Day 56

SECONDARY OUTCOMES:
To compare efficacy of a single IV application of FCM with that of placebo on change of iron status on Day 56 (i.e., proportion of subjects with haemoglobin (Hb) ≥12 g/dL; serum-ferritin (s-ferritin) ≥50 ng/mL; transferrin saturation (TfS) >20%). | Day 56
To determine the relationship between change in iron status (s-ferritin and TfS) and improvement of fatigue symptoms. | Day 56

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Favrat, Principal Investigator — Quartier UNIL-CHUV
Locations (1):
- Universitätsklinik für Frauenheilkunde, Vienna, Austria

REFERENCES:
- [Derived] Favrat B, Balck K, Breymann C, Hedenus M, Keller T, Mezzacasa A, Gasche C. Evaluation of a single dose of ferric carboxymaltose in fatigued, iron-deficient women--PREFER a randomized, placebo-controlled study. PLoS One. 2014 Apr 21;9(4):e94217. doi: 10.1371/journal.pone.0094217. eCollection 2014. PMID 24751822